CLINICAL TRIAL: NCT04101773
Title: Cost-effectiveness and Effectiveness of Rubber Band Ligation Versus Sutured Mucopexy Versus Haemorrhoidectomy in Patients With Recurrent Haemorrhoidal Disease: a Multicentre,Randomized Controlled Trial
Brief Title: Napoleon Trial: Optimal Treatment for Recurrent Haemorrhoidal Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 852002023
Record Dates: First submitted 2019-09-19; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Hemorrhoids
Keywords: hemorrhoids; haemorrhoidal disease; recurrence; rubber band ligation; haemorrhoidectomy
MeSH Terms: conditions — Hemorrhoids; Recurrence

STUDY DESIGN:
Intervention Model Description: Prospective multicentre randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: Due to the comparison of outpatient-based and surgical treatment strategies in this study, blinding to the treatment allocation for patients and medical staff is not possible. The trial statistician will be blinded for the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rubber Band Ligation (RBL) (Other): RBL is generallya simple, inexpensive procedure. It entails a ligation of haemorrhoids using rubber bands. In RBL, a disposable suction device applies a rubber band at least 2 cm proximal to the dentate line at the base of each haemorrhoidal cushion by using an anoscope. The banding process causes necrosis of the banded tissue and slough. The resultant inflammatory reaction causes refixation of the mucosa to the underlying tissue, helping to eliminate haemorrhoidal prolapse.The end result is a return of the haemorrhoidal cushions to a more normal size and configuration, with resolution of haemorrhoidal symptoms.
  Interventions: Procedure: RBL versus sutured mucopexy versus haemorrhoidectomy.
- Sutured mucopexy (Other): A sutured mucopexy is an operation performed under general anaesthesia. At 4 cm proximal of the dentate line, a Z- shaped stitch through the rectal wall is placed and then at the upper level of the haemorrhoidal tissue, pulling up the prolapsing haemorrhoid high into the anal canal.
  Interventions: Procedure: RBL versus sutured mucopexy versus haemorrhoidectomy.
- Haemorrhoidectomy (Other): Haemorrhoidectomy involves excision of the haemorrhoidal tissue. An elliptical incision is made in the external haemorrhoidal tissue extending proximally through the dentate line to the upper limit of the haemorrhoids. The base of the haemorrhoidal complex is ligated and the haemorrhoid is excised.
  Interventions: Procedure: RBL versus sutured mucopexy versus haemorrhoidectomy.

INTERVENTIONS:
Procedure: RBL versus sutured mucopexy versus haemorrhoidectomy. — All 3 interventions are part of Dutch usual care, and serve as each other's control.

SUMMARY:
Rationale: There is level I evidence in literature that the first management step of HD is basic treatment, including laxatives and high fibre dieti, ii. The next treatment modality after basic treatment in case of persistent symptoms is rubber band ligation (RBL), which can be repeated if necessary.

There is currently no consensus and a lack of evidence regarding the best treatment option for these patients having recurrent HD: continuing RBL or a surgical intervention. Furthermore, there is no estimate of costs and cost-effectiveness in this patient group.

Objective: The primary objective of this RCT is to compare the effectiveness of RBL, sutured mucopexy and haemorrhoidectomy regarding recurrence and patient-reported symptoms for recurrent grade 2 and 3 HD after at least 2 previous RBL treatments. Secondary objectives are to compare RBL, sutured mucopexy and haemorrhoidectomy for recurrent grade 2 and 3 HD after previous RBL treatments in terms of early and late complications, impact of symptoms on daily activities, patient satisfaction with treatment, health-related quality of life, costs and cost-effectiveness, and budget impact.

Study design: Dutch prospective multicentre randomized controlled trial.

Study population: Patients ≥18 who have recurrent grade 2 or 3 haemorrhoidal disease and who had at least 2 rubber band ligation treatments. In total, 558 patients will be included.

Intervention: Rubber band ligation versus sutured mucopexy versus haemorrhoidectomy. All three interventions are part of Dutch usual care, and serve as each other's control.

Main study parameters/endpoints: Primary outcomes are (1) recurrence and (2) patient-reported symptoms assessed after 12 months. Secondary outcome variables are early and late complications, impact of symptoms on daily activities, patient satisfaction with treatment, health-related quality of life, costs, cost-effectiveness and budget-impact.

DETAILED DESCRIPTION:
Haemorrhoidal disease (HD) is the most common type of anorectal complaint in the Netherlands, with an annual prevalence of 10% in general practice. There is level I evidence in literature that the first management step of HD is basic treatment,including laxatives and high fibre diet. The general practitioner usually offers basic treatment. If basic treatment fails patients are referred to the hospital. About 50.000 patients are referred to a hospital for HD in the Netherlands annually. The next treatment modality after basic treatment in case of persistent symptoms is rubber band ligation (RBL), which can be repeated if necessary. RBL is an easy, cheap and outpatient-based procedure. Thirty per cent of the patients, approximately 15.000 patients a year, develop recurrent symptoms after basic treatment and repeat RBL. There is currently no consensus and a lack of evidence regarding the best treatment option for these patients having recurrent HD: continuing RBL or a surgical intervention. Literature indicates that haemorrhoidectomy is the surgical treatment of choice based on outcomes like recurrencerate. The major drawback of this technique is that it is very painful and more costly compared to RBL. A relatively novel, but regular surgical alternative is the sutured mucopexy. Although hospital costs of sutured mucopexy are comparable to haemorrhoidectomy, the operation is less painful and requires less recuperation time. The recurrence rate of sutured mucopexy is ranked between that of RBL and haemorrhoidectomy.

A Dutch national survey conducted by our research group evaluating the management practices of HD demonstrated considerable variation in the best (surgical) treatment option regarding recurrent HD, resulting in potentially undesirable practice variation. The treatment of recurrent grade 2 or 3 HD currently depends on the preference and the experience of the surgeon and of the patient, without high level evidence substantiating this practice variation. This implies a need for a high quality study regarding the treatment of recurrent grade 2 or 3 HD. Diminishing this practice variation will endorse cost-effectiveness in healthcare settings.To our knowledge, this will be the first RCT worldwide comparing RBL, sutured mucopexy and haemorrhoidectomy in recurrent grade 2 or 3 HD and generating high-level evidence of the (cost-) effectiveness. The investigators consider combining 2 trials in one with a direct comparison between these three interventions to be an efficient research approach.

Up till now, trials were mostly powered on traditional outcomes like recurrence, a definition that differs widely between studies.To improve transparency between studies and facilitate the ability to compare and combine (future) studies, our research group developed a European Society of Coloproctology (ESCP) Core Outcome Set (COS) for HD. This international COS for HD selected 'patient-reported symptoms' as primary outcome. Additionally, the investigators recently developed a patient reported symptom score for HD: the PROM-HISS. This PROM is based on most cited symptoms in literature and patient interviews. The patient advisory board (PAB) of this project underlines the clinical relevance of this PROM. As the PROM-HISS has not yet been used in other studies and has to be validated, the investigators will additionally use patient-reported symptoms assessed by the PROM-HISS, next to recurrence, as primary outcome in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years or older
* Recurrent grade 2 or 3 HD
* Patients underwent at least 2 RBL treatments in the last 3 years based on hospital electronic patient file (EPD)
* Eligible for e-mail questionnaires
* Sufficient understanding of the Dutch written language (reading and writing)
* Obtained written informed consent

Exclusion Criteria:

* Previous rectal or anal surgery with the exception of rubber band ligation
* Patients that have had previous surgery treatment for HD (at any time)
* Previous rectal radiation
* Pre-existing sphincter injury
* Pathologies of the colon and rectum
* Medically unfit for surgery or for completion of the trial (ASA>III)
* Pregnancy
* Patients with hypercoagulability disorders
* Patients using Warfarin or Clopidogrel or oral anticoagulance therapy
* Patients that are unable to give full informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 558 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence | Assessed after 12 months post-intervention.
  The definition of recurrent HD is: "unchanged or worse symptoms of HD compared with before starting treatment".
Patient-reported symptoms measured with the PROM-HISS | The PROM-HISS will be completed by e-mail at four moments during follow-up: (1) at baseline; (2) 7 days; (3) 6 weeks; and (4) 12 months post-procedure.
  The Patient-Reported Outcome Measure-Haemorrhoidal Impact and Satisfaction Score (PROM-HISS) is a newly developed questionnaire assessing the symptoms of haemorrhoidal disease over time. These are blood loss, pain, prolapse, soiling and itching. These 5 items are graded using a 5-point Likert scale, ranging from (1) 'not at all', (2) 'a little', (3) 'reasonable', (4)'a lot' and (5) 'very much'. This results in a symptom score correlating with the severity of experienced HD symptoms. The PROM-HISS will be completed by e-mail. The PROM-HISS will assess a change of the symptoms over time. ThePROM-HISS is not validated yet, but an international validation study is being developed. Hence, the scale ranges are not clear yet.

SECONDARY OUTCOMES:
Early complication(s) - Abscess | This outcome measure will be assessed within 7 days post-procedure.
  Abscess will be assessed 7 days post-procedure. Abscess will be assessed by physical examination.
Impact of symptoms on daily life and patient satisfaction with treatment | The PROM-HISS will be completed by e-mail at four moments during follow-up: (1) at baseline; (2) 7 days; (3) 6 weeks; and (4) 12 months post-procedure.
  Assessed with the second part of the Patient-Reported Outcome Measure-Haemorrhoidal Impact and Satisfaction Score (PROM-HISS), which are each scored on a numeric rating scale from 0 to 10. Regarding impact of symptoms, 0 correlates with 'no impact at all' and 10 with 'highly impacted on daily life'. For patient satisfaction with treatment, this ranges between 0 'not satisfied' and 10 'very satisfied'. The PROM-HISS is not validated yet, but an international validation study is being developed. Hence, the scale ranges are not clear yet.
Health Related Quality of Life | The PROM-HISS will be completed by e-mail at four moments during follow-up: (1) at baseline; (2) 7 days; (3) 6 weeks; and (4) 12 months post-procedure.
  Measured by the EQ-5D-5L questionnaire and EQ-Visual Analogue Scale. These index scores are combined with length of life to calculate the QALY.
Early complication(s) - Urinary retention | This outcome measure will be assessed within 7 days post-procedure.
  Urinary retention will be assessed 7 days post-procedure. It will be assessed by ultrasonography.
Late complication(s) - Incontinence | Incontinence will be assessed at 52 weeks (1 year) post-procedure.
  The Wexner Fecal Incontinence Score will be used to assess incontinence.
Late complication(s) - Anal stenosis | Anal stenosis will be assessed at 52 weeks (1 year) post-procedure.
  Anal stenosis will be assessed by physical examination.
Late complication(s) - Fistula | Fistula will be assessed at 52 weeks (1 year) post-procedure.
  Fistula will be assessed by physical examination, in case this is inconclusive, MR imaging will be performed.
Costs | The questionnaires will be filled out at baseline, 6 weeks and 12 months follow-up.
  Total costs over the course of 12 months will be calculated by multiplying resource use with the costs per unit. Resource use(e.g. treatment, control visits, visits to the GP, other diagnostic/medical procedures, medication) will be obtained from the CRFand from recall cost-questionnaires (e.g. over the-counter medication, and lost work days). Sources for valuation of the costs will be cost prices of the Dutch costing manual and cost prices from thePharmaco therapeutic compass. If necessary, local hospital cost prices or otherwise NZa tariffs will be used, which are largely based on integral cost prices from the Dutch hospitals. Absence of work will be calculated by using the friction cost method,which is recommended by the Dutch manual for costing (Zorginstituut Nederland, 2015).
Cost-effectiveness | The EQ-5D-5L will be administered at baseline, 1 week, 6 weeks and at 12 months follow-up.
  The cost-effectiveness analysis from the healthcare perspective will be based on the cumulative proportion of patients whopresent with a recurrence up to 12 months follow-up. The cost-effectiveness analysis from the societal perspective (QALYs as outcome) will be based on the EQ-5D-5L.
Budget Impact Analysis | Time horizon of 5 years.
  A budget impact analysis (BIA) will be performed in accordance with the Dutch guidelines for economic evaluations and the ISPOR guidelines. The BIA will be performed from different perspectives (e.g. societal, healthcare) with a time horizon of 5 years. As input for the BIA, we will use the results that will become available from the clinical and cost-effectiveness study.The BIA will be performed using a simple decision analytic model. Different scenarios will be compared to investigate various levels of implementation or full substitution of any of the 3 interventions, as well as the swiftness of implementation (1-5 years). In order to test the robustness of the results, sensitivity analyses will be performed on data input and assumptions. No discounting will be performed. The target population in the BIA will be similar to the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Breukink, MD PhD, Study Chair — Maastricht University Medical Centre
Locations (16):
- Netherlands (16):
  - Maastricht University Medical Centre, Maastricht, Limburg
  - Ziekenhuisgroep Twente, Almelo
  - Meander Medisch Centrum, Amersfoort
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Gelre Ziekenhuizen, Apeldoorn
  - Rijnstate Ziekenhuis, Arnhem
  - IJsselland Ziekenhuis, Capelle aan den IJssel
  - Reinier de Graaf Gasthuis, Delft
  - Groene Hart Ziekenhuis, Gouda
  - Elkerliek Ziekenhuis, Helmond
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Laurentius Ziekenhuis, Roermond
  - Diakonessenhuis, Utrecht
  - Máxima Medisch Centrum, Veldhoven
  - VieCurie Medisch Centrum, Venlo

IPD SHARING:
Plan to Share IPD: Undecided
Not yet discussed with research group.

REFERENCES:
- [Derived] Kuiper SZ, Dirksen CD, Kimman ML, Van Kuijk SMJ, Van Tol RR, Muris JWM, Watson AJM, Maessen JMC, Melenhorst J, Breukink SO; Napoleon Trial Study Group. Effectiveness and cost-effectiveness of rubber band ligation versus sutured mucopexy versus haemorrhoidectomy in patients with recurrent haemorrhoidal disease (Napoleon trial): Study protocol for a multicentre randomized controlled trial. Contemp Clin Trials. 2020 Dec;99:106177. doi: 10.1016/j.cct.2020.106177. Epub 2020 Oct 17. PMID 33080380
- See also: ESCP Core Outcome Set for Haemorroidal Disease — https://www.escp.eu.com/images/guidelines/documents/ESCP-Core-Outcome_Set-for-haemorrhoidal-disease-Tol_et_al-2019-Colorectal_Disease.pdf
- See also: ESCP Guideline for Haemorroidal Disease — https://www.escp.eu.com/images/guidelines/documents/ESCP-Guidelines-Haemorrhoidal-Disease-2019-02.pdf